CLINICAL TRIAL: NCT06695013
Title: Immunobridging/Maintenance Therapy Versus Non-bridging Therapy in CAR-T Therapy for Low-risk Relapsed/Refractory B Cell Non-Hodgkin Lymphoma(R/R B-NHL): A Multicenter, Prospective, Randomized, Open-label, Controlled Clinical Study
Brief Title: Immunobridging/Maintenance Therapy Versus Non-bridging Therapy in CAR-T Therapy for Low-risk R/R B-NHL
Acronym: CART R/R NHL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLMB study
Record Dates: First submitted 2024-10-31; First posted 2024-11-19 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: B-NHL; CART Therapy
Keywords: Zanubrutinib; maintenance
MeSH Terms: interventions — zanubrutinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunotherapy bridging treatment (Experimental): Zanubrutinib ± radiotherapy was used as the bridging therapy in the immunobridging treatment group, a Follow-up maintenance treatment was determined according to the efficacy of D28 in the two groups. Patients with complete response (CR) were given no maintenance treatment, while patients with partial response (PR) were given Zanubrutinib orally plus PD-1 inhibitor for 2 years. Patients with stable SD or progressive PD were excluded from this study
  Interventions: Drug: zanubrutinib; Drug: CAR-T; Radiation: Bridging radiotherapy; Drug: Tislelizumab
- no bridging treatment (Active Comparator): The control group will not receive bridging treatment. Maintenance treatment will be consistent with the experimental group.
  Interventions: Drug: zanubrutinib; Drug: CAR-T; Drug: Tislelizumab

INTERVENTIONS:
Drug: zanubrutinib — zanubrutinib 160 mg BID orally
Drug: CAR-T — CAR-T Cell therapy
Radiation: Bridging radiotherapy — For patients in the experimental group, the decision regarding radiotherapy will depend on whether the specific lesions are suitable.
  Arms: Immunotherapy bridging treatment
Drug: Tislelizumab — 200mg IV Q3-4W

SUMMARY:
This study aims to explore whether adding immunotherapy bridging treatment for low-risk refractory/relapsed B-NHL can demonstrate better outcomes, in order to find the most effective treatment plan for low-risk patients.

DETAILED DESCRIPTION:
In the immunotherapy bridging treatment group, zanubrutinib ± radiotherapy will be used as the bridging treatment regimen, while those without bridging treatment will not receive bridging medications. Both groups will determine subsequent maintenance treatment based on efficacy at D28. Patients achieving complete response (CR) will not receive maintenance therapy, while those with partial response (PR) will be given oral zanubrutinib + PD-1 inhibitor for 2 years. Patients with stable disease (SD) or disease progression (PD) will not be included in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older, regardless of gender.
2. Histologically confirmed B-cell non-Hodgkin lymphoma, according to Lugano diagnostic criteria.
3. At least first-line treatment for relapsed or refractory patients, including chemotherapy regimens containing anthracyclines and anti-CD20 monoclonal antibody therapy; patients must meet definitions of refractory and recurrent.
4. No prior CD19 CAR T cell therapy.
5. Adequate organ function to assess tolerance to CAR-T therapy.
6. Sufficient vascular access for leukapheresis.
7. Ability to provide written informed consent and understand the study requirements and evaluation schedule.
8. Fertile patients must agree to use highly effective contraception during the study and for 120 days post-treatment.

Exclusion criteria：

Patients with any of the following conditions will not be included in the study:

1. History of allogeneic hematopoietic stem cell transplantation.
2. History of epilepsy, cerebrovascular ischemia/bleeding, dementia, cerebellar disease, or any autoimmune disease involving the central nervous system.
3. Any other malignancies within the past 2 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors (Ta, Tis, and T1).
4. Severe cardiovascular disease: NYHA grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias; NYHA grade III to IV heart failure or left ventricular ejection fraction (LVEF) < 50%.
5. Allergy to any investigational drug or excipient.
6. Active viral hepatitis requiring treatment, including chronic HBV carriers with HBV DNA ≥ 500 IU/mL and positive HCV RNA.
7. Active autoimmune disease or known history of allogeneic organ transplantation; long-term heavy use of immunosuppressants or other factors affecting study therapy.
8. Active infection.
9. History of uncontrolled systemic disease, such as diabetes or hypertension.
10. Known HIV infection.
11. Underlying medical condition or substance abuse that may interfere with drug administration or affect result interpretation, or increase treatment risk.
12. End-organ damage from autoimmune disease within the past 2 years or systemic use of immunosuppressive drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Complete response rate(CRR) at 3-month | 3 months post CAR-T infusion
  Complete response rate at 3-month is defined as the incidence of subjects achieving complete response (CR) at 3-month after CAR-T infusion according to the Lugano Classification, as determined by study investigators.

SECONDARY OUTCOMES:
Complete response rate(CRR) on D28 | 28 days post CAR-T infusion
  CRR on D28 after infusion is defined as the incidence of subjects achieving complete response (CR) on day 28 after CAR-T infusion according to the Lugano Classification, as determined by study investigators.
Objective remission rate (ORR) on D28 | 28 days post CAR-T infusion
  Objective remission rate (ORR) on D28 is defined as the incidence of either a CR or a partial response (PR) on day 28 after CAR-T infusion per the Lugano Classification as determined by study investigators.
Objective remission rate (ORR) at 3-month | 3 months post CAR-T infusion
  Objective remission rate (ORR) at 3-month is defined as the incidence of either a CR or a partial response (PR) at 3-month after CAR-T infusion per the Lugano Classification as determined by study investigators.
Progression-Free Survival (PFS) | 2 years post CAR-T infusion
  PFS is defined as the time from the CAR-T infusion date to the date of disease progression or death from any cause.
Overall Survival (OS) | 2 years post CAR-T infusion
  OS is defined as the time from CAR-T infusion to the date of death from any cause.
CAR-T cell expansion | 2 years post CAR-T infusion
  CAR-T cell expansion is to evaluate the proliferation and persistence of CAR-T cells in the patient's body following infusion. It is measured through quantitative assays, such as flow cytometry or qPCR, to track CAR-T cell levels in peripheral blood at predefined intervals.
Adverse Events rate | 2 years post CAR-T infusion
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin, Shanghai, Shanghai Municipality, China